CLINICAL TRIAL: NCT04931043
Title: Feasibility of Parent Training Using the Competent Learner Model With Families of Children With Autism Spectrum Disorder
Brief Title: Feasibility of Competent Learner Model With Families of Children With ASD
Status: Completed | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Jocelyn Stokes, Assistant Professor, West Virginia University
Other Study IDs: 1803052856
Record Dates: First submitted 2021-04-29; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Parent Training; Applied Behavior Analysis; Rural
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autism Spectrum Disorder (ASD) is a lifelong, neurodevelopmental disorder effecting one in fifty-nine children. Each individual with ASD is unique. Children with ASD may have trouble making friends, keeping friends, communicating their needs, engaging in leisure activities, learning to read and do math, and many other challenges. The children may engage in repetitive behaviors such as hitting themselves or flapping their hands, and may be over sensitive to particular sounds or lights which can make certain places, such as a store, very uncomfortable. Also, children with ASD may have challenging behaviors such as hitting others and excessive tantrums that can seem uncontrollable. 25 to 40 hours a week of intensive applied behavior analysis is the evidence-based treatment for children with ASD. Many children with ASD in rural areas and certain states are unable to access evidence-based treatment because of insurance barriers and lack of providers. The Competent Learner Model uses strategies from applied behavior analysis to target core skills that increase successful participation in life activities. Its program is applicable across all ages and developmental levels, and it has an online course of study which has been used to train professionals and lay people alike including parents. The purpose of this study was to assess the feasibility of training parents in applied behavior analysis using the Competent Learner Model with children with ASD who do not have access to treatment. The program consisted of a hybrid of group sessions for caregivers, coaching sessions for the caregiver-child dyads, and online units for caregivers. This project assessed participation in and satisfaction with the program as well as changes in parenting stress. Feedback from caregivers will be used to create a more satisfactory method of increasing accessing to families of children with Autism Spectrum Disorder in rural areas.

DETAILED DESCRIPTION:
Specific Aims: Many children with Autism in West Virginia are not able to access the evidence-based treatment, intensive applied behavior analysis, because of insurance barriers and lack of providers. Training parents in applied behavior analysis using the Competent Learner Model may allow children to access treatment. The purpose of this study was to determine if it is feasible to use online training units, group sessions for caregivers co-led by a parent, and family coaching sessions to improve the functioning of children with Autism. The current study is the first examination of Competent Learner Model as an independent intervention for parents using a hybrid of group and family sessions. Hypotheses: (1) Parent will complete therapy homework and attend 90% of sessions. (2) Parents will report a decrease in parenting stress.

Background: Autism is a lifelong, developmental disorder that affects 1 in 59 children, which represents about 720 children in the region of West Virginia where this study took place. Challenges for children with Autism include difficulty making and keeping friends, trouble talking to people, and insisting on rigid routines that interfere with daily life. The children may have challenging behavior such as hitting themselves, hitting others, and extreme meltdowns. Children may struggle to learn in typical classrooms, and may have trouble going to community events with their families. Families participate in fewer community activities leading to social isolation, and parents of children with Autism are more stressed than other parents. 25-40 hours per week of applied behavior analysis for 1-3 years is the evidence-based treatment for Autism. Many insurance companies in West Virginia specifically exclude services for children with Autism, and the Mountaineer Autism Project has estimated that only 1.6% of children with Autism in the state are receiving applied behavior analysis. Additionally, West Virginia has a limited number of providers for Autism. Children with Autism make greater progress across multiple settings (e.g., home, public) when their caregivers are involved in treatment, and coaching results in greater improvements in child behavior following behavioral parent training. Parent-implemented interventions for Autism are promising but more research is needed. When parents are trained to use the therapeutic strategies, the parent may be able to increase the child's skill development (e.g., self-care, functional academics, and social skills) across multiple settings and feel less stressed. The Competent Learner Model uses concepts and strategies from applied behavior analysis, Direct Instruction, and Precision Teaching to improve functioning of individuals with Autism. The program targets core skills that facilitate successful participation across all areas of an individuals' life, and it can be applied across all ages and developmental levels. A core component of the Competent Learner Model is the Course of Study, which has been used to train professionals and lay people. The Course of Study is a sequence of online training units using programmed instruction formats with embedded active student responding, video examples, and skill check outs. Coaching is a critical component of the program. While the Competent Learner Model uses well-researched strategies, the research of the program's effectiveness consists primarily of poster presentations and a handful of dissertations. One study found parents were better able to apply strategies and reported less stress when the parents were trained supplemental to their child's treatment. The effectiveness of the Competent Learner Model as implemented by parents independent of other treatment is unknown. Parent training using the Competent Learner Model may provide access to effective treatment for families. If this program is effective in training parents, it will increase access to effective services, decrease the amount of face-to-face time a parent must spend with a clinician and, thus, allow the clinician to serve a greater number of families simultaneously. More broadly, this treatment approach may present a treatment option for rural Americans with limited access to behavioral health outside of West Virginia as well. The study will contribute to the literature of training parents as therapists for their children with Autism.

ELIGIBILITY:
Inclusion Criteria: Caregiver-child dyads were eligible to participate if:

* the child has a diagnosis of Autism
* the child was under 18-years-old
* the child's legal guardian consented to treatment
* the child's insurance was accepted at this clinic or the family will pay for the services

Exclusion Criteria: Children were excluded from the study if:

* they were currently receiving intensive applied behavior analysis in the home
* the caregiver would not consent to being videotaped.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families were recruited through healthcare offices including primary care and behavioral health offices.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Session Attendance | Up to 16 weeks
  Number of sessions attended divided by total session
Homework Completion | Up to 16 weeks
  Number of training units completed in entirety divided by total units

SECONDARY OUTCOMES:
Parenting Stress Index Fourth Edition | From baseline to post intervention, up to 4 months
  36-item parent report questionnaire assessing stress in parent-child relationships, dysfunctional parenting, and child adjustment problems
Parent Sense of Competence Scale | From baseline to post intervention, up to 4 months
  Parent-report questionnaire assessing parenting attitudes and behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University Medicine University Behavioral Medicine and Psychiatry, Martinsburg, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Researchers may share data from the current study based on individual request from the other researcher

REFERENCES:
- [Background] Smith T, Iadarola S. Evidence Base Update for Autism Spectrum Disorder. J Clin Child Adolesc Psychol. 2015;44(6):897-922. doi: 10.1080/15374416.2015.1077448. PMID 26430947
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- [Background] McConachie H, Diggle T. Parent implemented early intervention for young children with autism spectrum disorder: a systematic review. J Eval Clin Pract. 2007 Feb;13(1):120-9. doi: 10.1111/j.1365-2753.2006.00674.x. PMID 17286734
- [Background] Stokes TF, Baer DM. An implicit technology of generalization. J Appl Behav Anal. 1977 Summer;10(2):349-67. doi: 10.1901/jaba.1977.10-349. PMID 16795561
- [Background] Baio J, Wiggins L, Christensen DL, Maenner MJ, Daniels J, Warren Z, Kurzius-Spencer M, Zahorodny W, Robinson Rosenberg C, White T, Durkin MS, Imm P, Nikolaou L, Yeargin-Allsopp M, Lee LC, Harrington R, Lopez M, Fitzgerald RT, Hewitt A, Pettygrove S, Constantino JN, Vehorn A, Shenouda J, Hall-Lande J, Van Naarden Braun K, Dowling NF. Prevalence of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2014. MMWR Surveill Summ. 2018 Apr 27;67(6):1-23. doi: 10.15585/mmwr.ss6706a1. PMID 29701730
- [Background] Mancil G. R., Boyd, B. A., & Bedersem, P. Parental stress and autism: Are there useful coping strategies? Education and Training in Developmental Disabilities. 2009; 44:4; 523-537.
- [Background] Burrell, T. L., & Borrego, J. Parents' involvement in ASD treatment: What is their role? Cognitive and Behavioral Practice. 2012; 19(3): 423-432.
- [Background] Tucci, V., Hursh, D., Laitinen, R., & Lambe, A. Competent learner model for individuals with autism/ PDD. Exceptionality. 2005; 13(1); 55-63.
- [Background] Lofton, K. L. Autism services lacking for West Virginia families. Appalachia Health News. April 6, 2016. wvpublic.org/post/autism-services-lacking-west-virginia-families. Accessed March 5, 2018.